CLINICAL TRIAL: NCT06285682
Title: The Dose Response of a Commercially Available Olive Fruit Water (OliPhenolia®) on the Bioavailability of Hydroxytyrosol, and Its Metabolites, Over a Four-hour Time Period in Healthy Adult Humans.
Brief Title: Bioavailability of Hydroxytyrosol in Healthy Adult Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Anglia Ruskin University (Other)
Collaborators: Fattoria La Vialla (Unknown); Instituto Kurz (Unknown)
Responsible Party: Principal Investigator, Justin Roberts, Professor, Anglia Ruskin University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: ETH2324-2826
Record Dates: First submitted 2024-02-23; First posted 2024-02-29 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Healthy
Keywords: Hydroxytyrosol; Bioavailability

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned a dose of olive-derived hydroxytyrosol in a double-blind manner. Following a ≥3 day wash out participants then cross-over to an alternate dose. This process is then repeated for the third and final dose.
Who Masked: Participant, Investigator
Masking Description: Volume of nutritional supplement is provided in a double-blinded manner. Both participants and research testers will be masked from knowing the specifics of the volume allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- 0.5mg∙kg-1 olive derived hydroxytyrosol from OliPhenolia®. (Experimental): Olive derived hydroxytyrosol will be ingested via a commercially available olive fruit wastewater (OliPhenolia®) in a dose relative to participant body mass. In this arm participants will consume and oral bolus of 0.5mg∙kg-1 olive derived hydroxytyrosol.
  Interventions: Dietary Supplement: OliPhenolia®)
- 1.0mg∙kg-1 olive derived hydroxytyrosol from OliPhenolia®. (Experimental): Olive derived hydroxytyrosol will be ingested via a commercially available olive fruit wastewater (OliPhenolia®) in a dose relative to participant body mass. In this arm participants will consume and oral bolus of 1.0mg∙kg-1 olive derived hydroxytyrosol.
  Interventions: Dietary Supplement: OliPhenolia®)
- 1.5mg∙kg-1 olive derived hydroxytyrosol from OliPhenolia®. (Experimental): Olive derived hydroxytyrosol will be ingested via a commercially available olive fruit wastewater (OliPhenolia®) in a dose relative to participant body mass. In this arm participants will consume and oral bolus of 1.5mg∙kg-1 olive derived hydroxytyrosol.
  Interventions: Dietary Supplement: OliPhenolia®)

INTERVENTIONS:
Dietary Supplement: OliPhenolia®) — Olive derived hydroxytyrosol will be ingested via a commercially available olive fruit wastewater (OliPhenolia®) in a dose relative to participant body mass. Participants will consume three doses within the entire study, one dose per visit, separated by a ≥3 day wash out period.

SUMMARY:
Brief summary: There is current scientific interest in hydroxytyrosol due to its anti-inflammatory and antioxidant properties, efficient protection of vascular tissue and ability to neutralise free radicals via hydrogen donation. Recognised as the potent polyphenol within a commercially available olive-fruit water (OliPhenolia®), data from this research will determine the dose of OliPhenolia® required for the optimum absorption and metabolism of hydroxytyrosol. The primary aim of this research is to identify the dose of hydroxytyrosol (0.5, 1.0 or 1.5 mg∙kg-1) within OliPhenolia® that demonstrates the greatest area under the plasma concentration curve for hydroxytyrosol over a four-hour period. A secondary aim is to assess maximum concentration (CMAX) and time to maximum concentration (TMAX) of total hydroxytyrosol and secondary metabolites (Tyrosol, HT-3-glucoronide, HT-3-sulphate, 3,4-Dihydroxyphenylacetic Acid, Homovanillic Acid and Oleuropein) following consumption of 3 randomised doses of OliPhenolia® on separate occasions with healthy adult volunteers.

DETAILED DESCRIPTION:
There is current and significant scientific interest in the use of plant-based polyphenol supplementation to support health, protection against disease and recovery from exercise. Recent literature dictates that daily supplementation (~3d of >1,000mg of polyphenols) may enhance recovery from exercise and can therefore be associated with both an increased frequency of exercise and quality of movement. The large proportion of research to date has focussed on certain fruit extracts (blackcurrant, tart Montmorency cherry or pomegranate juice), however a recent study from our group utilising milled waste olive-water demonstrated that 16 days of supplementation may support recovery from exercise via the blunting of certain oxidative stress markers and enhance low-intensity exercise performance through a reduction in oxygen economy.

To date there has been significant clinical research interest in the properties of waste-water produced when cold pressing olives, which has been shown to contain high concentrations of natural polyphenols, particularly hydroxytyrosol, a potent scavenger of free radicals. Fattoria La Vialla is an Italian-based organic farm producing various products including cold-pressed olive oil. In doing so, they also produce an olive waste-water extract which is commercially available as 'OliPhenolia®' and currently advertised as a 'health promoting supplement'. Whilst several clinical studies have been undertaken using this product, to date there have been no studies investigating the dose response of OliPhenolia® on the bioavailability of hydroxytyrosol, and the secondary metabolites. As such this study proposes to investigate the bioavailability of hydroxytyrosol across three doses of OliPhenolia® (0.5, 1.0 or 1.5mg∙kg-1) in a randomised manner to understand and therefore inform pertinent supplementation strategies to support health and components of exercise.

Following a study briefing and provision of written informed consent, participants will be required to attend the Human Physiology Laboratory at Cambridge Centre for Sport and Exercise Sciences, Anglia Ruskin University on three occasions. Each visit will follow an identical protocol, providing an randomly assigned dose (0.5, 1.0 or 1.5mg∙kg-1) of olive derived hydroxytyrosol from OliPhenolia® (based on body weight). Participants will be required to complete a weighed food diary and adhere to a 'low-polyphenol' diet for the three days prior to each visit, as well as consume a standardised pre-visit evening meal the night before each visit. Participants will arrive at each visit in a fasted (~10h) and hydrated state (500mL 1h prior to arrival). Following a resting blood sample, participants will consume one of the three doses of OliPhenolia® and then remain in a comfortable supine position for the remainder of the visit. Water will be provided at 90 and 180 minutes post OliPhenolia® consumption.

Blood samples - two 4mL wholeblood samples will be collected via cannulation at rest and then 20,40, 60, 120 and 240 minutes following each dose. Following collection, blood samples will be immediately centrifuged with plasma allocated into separate cryovials pre treated with 150µL citric acid for the analysis of: i) the main polyphenol compound- hydroxytyrosol; ii) the secondary metabolites of hydroxytyrosol (Tyrosol, HT-3-glucoronide, HT-3-sulphate, 3,4-Dihydroxyphenylacetic Acid, Homovanillic Acid and Oleuropein).

Nutritional supplementation - all products will be supplied/certified independently via Fattoria La Vialla, Italy (https://www.oliphenolia.it/uk/).

ELIGIBILITY:
Inclusion Criteria:

* UK based men and women aged ≥ 21 - 65
* Written, witnessed and cosigned informed consent
* Willingness and ability to conform to the full protocol

Exclusion Criteria:

* Current or recent (within the last 4 weeks) engagement with a strict dietary regime i.e., vegetarian / vegan / ketogenic / paleolithic / high protein / weight loss.
* Any known issues with blood taking.
* Any known bleeding disorders.
* Any known allergy to olives, grapes or prunes.
* Average alcohol use of >21 glasses per week for men and >14 glasses per week for women (on average for the last six months).
* Any drug or medicine abuse in the last six months
* Known cardiovascular disease, disease related to the immune system (including HIVand hepatitis) and / or the respiratory system.
* Known Diabetes Mellitus type I or type II.
* Known renal or liver issues or known thyroid dysfunction.
* Currently undertaking regular heavy and / or extreme exercise (please discuss with the lead researcher if you are unsure).
* Current smoker or stopped smoking for <one month prior to the first visit.
* Major medical or surgical event requiring hospitalisation in the previous three months and / or any scheduled during the scheduled study period.
* Current participation in any other clinical study within the month previous to the study start date (discuss with the lead researcher if unsure).
* Known pregnancy and / or lactation (women only)

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2024-02-03 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Hydroxytyrosol bioavailability | Four hours
  Area under the plasma concentration curve of hydroxytyrosol (mg/L)
Bioavailability of hydroxytyrosol metabolites. | Four hours
  Area under the plasma concentration curve of Tyrosol, HT-3-glucoronide, HT-3-sulphate, 3,4-Dihydroxyphenylacetic Acid, Homovanillic Acid and Oleuropein (mg/L)

SECONDARY OUTCOMES:
Hydroxytyrosol CMax | Four hours
  Hydroxytyrosol peak plasma concentration (CMAX) in mg/L
Hydroxytyrosol TMAX | Four hours
  Time to peak hydroxytyrosol (TMAX in minutes) - hydroxytyrosol measured in mg/L
CMAX of hydroxytyrosol secondary metabolites | Four hours
  Peak plasma concentration (CMAX) of Tyrosol, HT-3-glucoronide, HT-3-sulphate, 3,4-Dihydroxyphenylacetic Acid, Homovanillic Acid and Oleuropein - all measured in mg/L
TMAX of hydroxytyrosol secondary metabolites | Four hours
  Time to peak concentration (TMAX in minutes) of Tyrosol, HT-3-glucoronide, HT-3-sulphate, 3,4-Dihydroxyphenylacetic Acid, Homovanillic Acid and Oleuropein - all metabolites measured in mg/L

CONTACTS AND LOCATIONS:
Overall Officials: Justin D Roberts, PhD, Principal Investigator — Anglia Ruskin University
Locations (1):
- Cambridge Centre for Sport and Exercise Sciences, Anglia Ruskin University, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: No